CLINICAL TRIAL: NCT03087123
Title: Physical and Social Environmental Influence on Children's Exercise: Preparation (Pre-PLACE)
Acronym: Pre-PLACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Stephanie Broyles, Associate Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: PBRC 2016-068
Record Dates: First submitted 2017-03-15; First posted 2017-03-22 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Physical Activity
Keywords: single-case design; children; health equity; mobile health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: In accordance with a single case design approach, where each subject acts as his/her own control, families will be randomized to a 2, 4, or 6-week baseline period before being administered the P-Mobile app based intervention. All families will receive the same P-Mobile intervention following the baseline period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2-Week Baseline (Active Comparator): Families will be randomized to a 2-week baseline period before being administered the P-Mobile app based intervention. All families will receive the same P-Mobile intervention following the baseline period. The intervention will consist of 10 lessons delivered over 12 weeks designed to increase physical activity in children. The lessons will be delivered weekly and are the same ones utilized in the P-Mobile pilot study. The parents will also receive notifications designed to prompt physical activity, motivate, and remind parents of lesson content.
  Interventions: Behavioral: P-Mobile App
- 4-Week Baseline (Active Comparator): Families will be randomized to a 4-week baseline period before being administered the P-Mobile app based intervention. All families will receive the same P-Mobile intervention following the baseline period. The intervention will consist of 10 lessons delivered over 12 weeks designed to increase physical activity in children. The lessons will be delivered weekly and are the same ones utilized in the P-Mobile pilot study. The parents will also receive notifications designed to prompt physical activity, motivate, and remind parents of lesson content.
  Interventions: Behavioral: P-Mobile App
- 6-Week Baseline (Active Comparator): Families will be randomized to a 6-week baseline period before being administered the P-Mobile app based intervention. All families will receive the same P-Mobile intervention following the baseline period. The intervention will consist of 10 lessons delivered over 12 weeks designed to increase physical activity in children. The lessons will be delivered weekly and are the same ones utilized in the P-Mobile pilot study. The parents will also receive notifications designed to prompt physical activity, motivate, and remind parents of lesson content.
  Interventions: Behavioral: P-Mobile App

INTERVENTIONS:
Behavioral: P-Mobile App — The behavioral strategies are based on Social Cognitive Theory. The following topics will be covered: self-monitoring, goal setting, stimulus control, making time for exercise, exercising in- and outdoors, problem-solving, reinforcing PA, reducing sedentary behaviors, relapse prevention, parental modeling, lifestyle exercise, self-efficacy, self-management, parental PA modeling, parental co-participation, and establishing PA rules. Parents will be provided with adapted step goals (based on principles of shaping). Text messages will be designed to prompt PA, remind parents of concepts from the lessons, and motivate behavioral change.

SUMMARY:
Community based interventions are more acceptable to community members when all participants receive the intervention. A 'stepped-wedge' or 'multiple-baseline' design allows for all participants to receive the intervention by randomizing participants into conditions defined by the length of the baseline period. The primary aim of this pilot study is to gather data that will allow the researchers to estimate parameters, such as the appropriate length of the baseline period that will allow them to power a larger study. A second key aim is to determine if a smartphone intervention that is delivered to parents can increase physical activity in their 6-10 year old inactive children.

DETAILED DESCRIPTION:
Low levels of physical activity in childhood are related to obesity and risk for diabetes and cardiovascular disease. This translational study is an attempt to take interventions that have been shown to be effective in highly controlled setting and implement them in the community. We will utilize a form of a single case design (i.e., stepped-wedge or multiple-baseline design), which is an underused, though promising, alternative to the traditional, parallel-group randomized trial in which each study participant acts as his/her own control. Participants will be randomized to baseline periods of varying length such that the change in the study outcome can be causally attributed to introduction of the intervention. In accordance, families will be randomized to a 2, 4, or 6-week baseline period before being administered the P-Mobile app based intervention. All families will receive the same P-Mobile intervention following the baseline period. The P-Mobile intervention will be delivered to parents via the P-Mobile smartphone app; it consists of 10 lessons designed to increase physical activity in children. The parents will also receive notifications designed to prompt physical activity, motivate, and remind parents of lesson content. The intervention will also utilize an adaptive step goal approach, in which the step goal is modified based on each participant's individual performance. The primary aims of the study are: (1) To estimate several parameters, which will allow us to redesign our study as a single case design (and to conduct simulation-based power calculations): (a) average day-to-day variability in daily steps during the baseline period, (b) average autocorrelation in the daily step data, and (c) average effect size at 2 weeks, 4 weeks, and 6 weeks after introduction of the intervention. (2) To test the feasibility of the P-Mobile app (3) To demonstrate our ability to recruit participants from targeted neighborhoods.

ELIGIBILITY:
Inclusion Criteria:

The child must:

* Be 6-10 years of age
* Have at least one participating parent.
* Be Physically capable of exercise
* Have an average steps/day less than the 50th percentile for age and gender (e.g., <8,900 steps/day for 10-year old girls and <10,200 steps/day for 10-year old boys).

The parent must:

* Have a smartphone
* Be willing to download and use the P-Mobile app
* Demonstrate the ability to send text messages
* Have no plans to move during the study period (up to 4 months)

Families must:

•Reside in targeted geographic area

Exclusion Criteria:

Exclusion criteria for the child includes:

* Significant cardiovascular disease or disorders via self-report
* Other significant medical problems that would prevent them from engaging in regular physical activity.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Physical activity | Baseline.
  Fitbit®: The child will wear a wireless activity monitor (Fitbit®) for the entire study. The Charge 2 wrist-worn Fitbit will be utilized.

SECONDARY OUTCOMES:
Height | Baseline, Week 4, 8, and 12.
  Height will be measured using a standard stadiometer and will be measured to the nearest 0.1 kg
Weight | Baseline, Week 4, 8, and 12.
  Weight will be measured using a balance beam scale without shoes and will be recorded to the nearest 0.1 cm.
Body composition | Baseline, Week 4, 8, and 12.
  The Tanita Body Composition Analyzer (model TBF-310) will be used to measure body weight and impedance (a measure of body fat and lean muscle mass).
Home and neighborhood environment questionnaire | Baseline, Week 4, 8, and 12.
  Parents will report their perceptions of the neighborhood social environment, the neighborhood built and physical activity environment, and the home food and physical activity environment.
Sibling Relationship Inventory (SRI). | Baseline, Week 4, 8, and 12.
  Participants will be asked to complete the Sibling Relationship Inventory. The SRI is intended to evaluate the participant's relationship with the child closest in age and currently living in the participant's household.
Treatment satisfaction | Week 12
  This 15-item questionnaire assesses parents' satisfaction with the intervention in four domains 1) Overall Satisfaction, 2) Helpfulness, 3) Ease of Use, and 4) Perceived Change in Physical Activity.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Broyles, Ph.D., Principal Investigator — Pennington Biomedical Research Center; Robert L. Newton, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No